CLINICAL TRIAL: NCT07263789
Title: Randomized, Open-label, Parallel Group Study to Evaluate the Efficacy of Euglycem in Reducing Blood Glucose in Patients With Dysglycemia After Three Months of Treatment - EUGLYCARE Study
Brief Title: Effect of a Food Supplement on Blood Glucose Levels in Patients With Impaired Glucose Values
Acronym: EUGLYCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Giuseppe Derosa, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EUGLYCARE
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Dysglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Euglycem (Active Comparator): An association of banaba leaves extract and chromium picolinate
  Interventions: Dietary Supplement: Nutraceutical supplements
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutraceutical supplements — An association of banaba leaves extract and chromium picolinate (Euglycem®) will be administered
  Arms: Euglycem
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the efficacy of Euglycem® plus recommended standard diet on reducing FPG compared to baseline and to recommended standard diet alone after 3 months

DETAILED DESCRIPTION:
Dysglycemia (or prediabetes) is a reversible metabolic condition that increases the risk of developing type 2 diabetes mellitus, a pathological condition that, in prognostic terms, is considered equivalent to cardiovascular disease. Type 2 diabetes mellitus, therefore, is a serious pathology not only for the symptoms and complications related to it but also for the prognosis. Dysglycemia is characterized by an alteration in blood glucose levels that do not yet fall within the diagnostic criteria for diabetes. It is a very common condition that often remains unknown because it is asymptomatic. Dysglycemia is due to a receptor dysregulation between cellular and circulating glucose values and pancreatic insulin production, characterized by an initial resistance to insulin produced by pancreatic beta cells and directed to the muscle cells. Insulin acts as a catalyst for the use of glucose for metabolic purposes with consequent withdrawal of circulating glucose and, therefore, reduction of glycemia. If this regulation does not work perfectly, blood glucose levels increase and the condition of dysglycemia is feared. The main risk factors associated with dysglycemia are overweight and obesity, family history of diabetes, sedentary lifestyle, hypertension and hypercholesterolemia, all risk factors also for cardiovascular diseases. In women dysglycemia is often also correlated with polycystic ovary and gestational diabetes. There is evidence that dysglycemia and type 2 diabetes are associated with a deficiency of vitamin D. The pancreatic beta cells, responsible for the release of insulin, express receptors for vitamin D and their dysfunction is demonstrated in various experimental models. However, the administration of vitamin D to subjects with dysglycemia or diabetes has produced uncertain results. Dysglycemia is a silent condition, therefore asymptomatic, although subjects with dysglycemia are, in general, already exposed to an increased risk of developing cardiovascular diseases. Consequentially, the diagnosis is exclusively laboratory, i.e. a fasting blood glucose (FPG) between 100 and 125 mg/dl, a glucose load curve (OGTT) whose result after two hours is higher than 140 mg/dl (normal limit) and less than 200 mg/dl (diagnostic criterion for type 2 diabetes mellitus), i.e. between 140-199 mg/dl and glycated hemoglobin (HbA1c) values between 5.7-6.4%. It is believed that approximately 11% of subjects with dysglycemia develop type 2 diabetes after three years. This percentage rises to 25% after five years. The remedies to overcome the prediabetic condition are essentially based on the reduction of risk factors and relative improvement of lifestyle. A healthy diet, low in fat and rich in fiber and vegetable protein is important together with physical activity to be practiced according to World Health Organization (WHO) recommendations. To date, no drug is approved for the treatment of dysglycemia, while substances of natural origin have been shown to contribute to the normalization of glucose metabolism in association with the above mentioned remedies which are known to present long-term compliance problems. This is the context in which the association of banaba leaves extract and chromium picolinate (Euglycem®) is positioned. Chromium is an essential mineral that improves insulin sensitivity. It also has favorable effects on the metabolism of proteins, carbohydrates and fats and leads to a reduction in body weight. Chromium deficiency is rare, but significant, because it results in poorer glycemia and cholesterolemia control. Banaba leaves extract promotes the absorption of glucose and its use for energy purposes, thus playing a role in the regulation of blood glucose and insulin levels. By regulating glycemia fluctuations that activate the hunger center, banaba is useful for reducing body weight and triglyceride levels. One study reported that in 10 healthy subjects who received 1 tablet/day of Euglycem containing 50 mg of banaba leaves extract or placebo for 4 days, the supplement significantly reduced the glucose area under the curve (AUC) and insulinemia after glucose load compared to placebo. The same study also evaluated the effect of the supplement in 40 subjects with dysglycemia randomized to receive 1 tablet/day of Euglycem containing 10 mg or 50 mg of banaba leaves extract for 4 weeks associated with an improvement in dietary and behavioral habits. It was highlighted that both dosages improved weight, body mass index (BMI), FPG and Homeostasis Model Assessment (HOMA) index compared to baseline while only the highest dose significantly reduced fasting plasma insulin (FPI) and HbA1c compared to baseline. However, the study has important limitations such as the small number of subjects enrolled and the short duration of treatment.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤30 kg/m2
* subjects able to understand the informed consent and sign it before enrollment in the study
* subjects willing to follow all study requirements and perform all study visits as well as collaborate with the investigator.

Exclusion Criteria:

* ongoing treatment with drugs that can affect blood glucose
* current participation in another investigational drug or investigational device trial or inclusion in another investigational drug or investigational device trial within the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Dysglicemia | 3 months
  The primary objective is to evaluate the efficacy of Euglycem® plus recommended standard diet on reducing FPG compared to baseline and to recommended standard diet alone after 3 months of supplementation.

SECONDARY OUTCOMES:
Insulin reistance | 3 months
  The secondary objective is to evaluate the efficacy of Euglycem® plus recommended standard diet on reducing HbA1c, FPI and HOMA index
Vitamin D3 levels | 3 months
  The secondary objective is to evaluate the efficacy of Euglycem® plus recommended standard diet on the variation of vitamin D3 levels
Glycemic status | 3 months
  The secondary objective is to evaluate the efficacy of Euglycem® plus recommended standard diet on the proportion of subjects pass from impaired fasting glycemia (IFG) condition to euglycemia and the proportion of subjects pass from impaired glucose tolerance (IGT) condition to euglycemia

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Policlinico San Matteo, Pavia, Lombardy
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia

IPD SHARING:
Plan to Share IPD: No